CLINICAL TRIAL: NCT01305837
Title: Cyclic Oral Methylprednisolone Trial in Multiple Sclerosis
Acronym: COMTiMS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Rikke Ratzer, MD, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2010-370; 2010-024561-43 (EudraCT Number)
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2013-07-11 (Estimated); Status verified 2013-07

CONDITIONS: Progressive Multiple Sclerosis
Keywords: multiple sclerosis; methylprednisolone; osteopontin; inflammation; demyelinating
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis; Inflammation | interventions — Methylprednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- methylprednisolone (Experimental): all patients will be treated with the active drug methylprednisolone 500 mg in 3 days every month for 60 weeks.
  Interventions: Drug: methylprednisolone

INTERVENTIONS:
Drug: methylprednisolone — 500 mg of methylprednisolone taken in 3 days every month
  Other Names: Medrol

SUMMARY:
The purpose of this study is to determine whether cyclic oral methylprednisolone once every month has an effect on the intrathecal inflammation in patients suffering from progressive multiple sclerosis.

DETAILED DESCRIPTION:
Multiple Sclerosis (MS) is a chronic inflammatory demyelinating disease of the central nervous system (CNS). It is presumably T-cell mediated and it is the most common non-traumatic cause of disability affecting young people. 85 % of the MS causes starts out as relapsing remitting MS (RRMS) and 15 % as primary progressive MS (PPMS). It has been found that after 10 years 40-45 % of the RRMS patients will convert to a more progressive state of disease, secondary progressive MS (SPMS).

Until recently it has been believed that the progression seen in MS occurred because of axonal loss and neurodegeneration could occur independently of inflammation. Now neuropathology studies shows that there is a close association between inflammation and neurodegeneration in all stages of MS - also the progressive forms of MS.

Osteopontin (OPN) is an extracellular matrix protein with chemokine, cytokine and intergrin properties. It has multiple immunological functions and is secreted by activated macrophages, leukocytes and activated T lymphocytes. It is present in extracellular fluids and is up-regulated at sites of inflammation. Increased levels of OPN where reported in the cerebrospinal fluid (CSF) in patients with MS.

The main aim of this study is to analyze the effect of cyclic oral methylprednisolone on the intrathecal inflammation in patients suffering from progressive multiple sclerosis measured by OPN in the CSF. Second the investigators will look at other aims of intrathecal inflammation, neurodegeneration, demyelination and safety.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years old
* Progressive form of MS (Eg. primary or secondary progressive MS)
* Duration of progressive phase at least 1 year
* Progression of at least 1 EDSS point for the last 2 years or at least ½ EDSS point in patients with EDSS > 5,5
* Progressin in 2 FS point
* EDSS </= 6,5
* Signed informed consent and written authority

Exclusion Criteria:

* Pregnancy and breast feeding
* Lack of secure contraception for women of child-bearing age (hormonal or intrauterine device)
* Attack in the last month previous to inclusion
* Treatment with methylprednisolone or cyclic methylprednisolone the 3 previous month before inclusion
* Treatment with interferon-beta, Glatiramer acetate, immunglobulin G or other immunomodulating treatment the 3 previous month before inclusion
* Treatment with Mitoxantrone, ciclofosfamide, Azathioprin or other immunosuppressive treatment the 6 previous month before inclusion
* Previous treatment with drugs which the treating physician finds could have influence on the study results
* Diseases associated with immune defects
* Treatment with other anticoagulant than acetyl salicyl acid
* Malignancy
* Diabetes Mellitus
* Renal insufficiency or S-Creatinine > 150 mmol/l
* Acute or chronic infections with hepatitis B og C virus, HIV or other infections which the treating physician finds relevant
* Psychiatric illness or other conditions which can impair the collaboration of the patient participating in the study
* Contra-indication to MRI
* Hypersensitivity to methylprednisolone
* Osteoporosis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-04; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
CSF osteopontin | baseline and week 60

SECONDARY OUTCOMES:
aims for clinical progression | baseline and week 60
  1. Change in expanded disability status scale (EDSS)
  2. Change in Timed 25-foot Walk (T25FW)
  3. Change in Multiple sclerosis impairment scale (MSIS)
  4. Change in multiple sclerosis functional composite (MSFC)
  5. Change in short form 36 (SF-36)
aims for demyelination and disease activity | baseline, week 12 (only MRI aims and MEP) and week 60
  1. Change in the concentration of neurofilament heavy chain (NfH) in CSF 2. Change in the concentration of myelin basic protein (MBP) i CSF 3. Change in normalised brain volume (NBV), grey matter volume (GMV) og white matter volume (WMV) 4. Change in MTR og DTI i hele hjernen, lesions, normal appearing grey matter (NAGM) og normal appearing white matter (NAWM) 5. MEP (motor evoked potentials)
aims of intrathecal inflammation | baseline and week 60
  1. Change in cellcount i CSF
  2. Change in IgG-index
  3. Change in the concentration of nitric oxid (NO) metabolittes in CSV
  4. Change in CSV-serum albumin qvotient
  5. Change in the concentration of CXCL13 i CSF
  6. Change in the concentration of MMP-9 i CSF
  7. Number of new Gd-enhancing lessions on MRI
  8. Volume of T2 lessions on MRI
  9. Number of new or bigger T2 lessions on
  10. Change in MTR in the hole brain, in lessions, grey matter og white matter
  11. Change in DTI the hole brain, in lessions, grey matter og white matter
safety | screnning, baseline, week 12, 24, 36, 48, 60
  physical examination, blood pressure, pulse, DEXA scan, bloodtests

CONTACTS AND LOCATIONS:
Overall Officials: Rikke Ratzer, MD, Principal Investigator — Scleroseklinikken, Rigshospitalet; Per S Sørensen, Professor, MD, Study Chair — Scleroseklinikken, Rigshospitalet
Locations (1):
- Scleroseklinikken, Rigshospitalet, Copenhagen, Denmark